CLINICAL TRIAL: NCT06593990
Title: Left Atrial Function and Dimensions As Predictors of Disease Activity in Rheumatoid Arthritis Patients
Brief Title: LA Function and Dimensions As Predictors of Disease Activity in RA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohammed ragab, Assistant lecturer in assiut university, Assiut University
Other Study IDs: Left atrial function in RA
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rhematoid Arthritis
Keywords: left atrial function; rhematoid arthritis; musculoskeletal ultrasound; echocardiographic changes in rhematoid arthritis
MeSH Terms: interventions — Blood Cell Count; Blood Sedimentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: echocardography — Patients will be subjected to transthoracic echocardiography including, the following parameters will be measured:
  * Left ventricular (LV) dimensions: end diastolic and systolic dimensions and LV ejection fraction (EF).
  * Trans- mitral Doppler flow velocities including early (E) and late(A) diastolic velocities, E/A ratio.
  * LA anteroposterior diameter measure from 2D parasternal long axis view targeted M-mode.
  * LA superior-inferior and medio-lateral diameters measure from the apical 4 chamber view.
  * LA volume included:
  * Maximal LA volume measure at the end of systole
  * Minimal LA volume will be measured at end diastole just at the closure of the mitral valve.
  * Pre contractile LA volume ( LAV pre-A] measured at P-wave onset on ECG just before atrial contraction.
  Other Names: musculoskeletal ultrasound
Device: musculoskeletal ultrasonography — Ultrasound detected synovitis t
Diagnostic Test: lipid profile test — The lipid profile typically includes measurement of total cholesterol, HDL-cholesterol (often called good cholesterol), LDL-cholesterol (often called bad cholesterol), and triglycerides.
Diagnostic Test: C reactive protein — A c-reactive protein test measures the level of c-reactive protein (CRP) in a sample of your blood. CRP is a protein that your liver makes. Normally, you have low levels of c-reactive protein in your blood. Your liver releases more CRP into your bloodstream if you have inflammation in your body. High levels of CRP may mean you have a serious health condition that causes inflammation.
Diagnostic Test: Complete blood count CBC — A complete blood count, or CBC, is a blood test that measures many different parts and features of your blood, including:
  Red blood cells, which carry oxygen from your lungs to the rest of your body. White blood cells, which fight infections and other diseases. There are five major types of white blood cells. A CBC test measures the total number of white cells in your blood. A different test called a CBC with differential measures the number of each type of these white blood cells.
  Platelets, which stop bleeding by helping your blood to clot. Hemoglobin, a protein in red blood cells that carries oxygen from your lungs to the rest of your body.
  Hematocrit, a measurement of how much of your blood is made up of red blood cells.
  Mean corpuscular volume (MCV), a measure of the average size of your red blood cells.
Diagnostic Test: Erythrocyte sedimentation rate (ESR). — An erythrocyte sedimentation rate (ESR) is a blood test that that can show if you have inflammation in your body. Inflammation is your immune system's response to injury, infection, and many types of conditions, including immune system disorders, certain cancers, and blood disorders.
Device: x ray of the hand — The X-ray may show a hand with advanced rheumatoid arthritis. "Bone erosion" means cartilage and bone are worn away. "Bone displacement" means that a bone has moved out of its normal position. This X-ray shows how bone erosion and bone displacement can change the shape of the hand.

SUMMARY:
the aim of this study is to

* describe subclinical echocardiographic changes of the LA (dimensions and function) in patients with rheumatoid arthritis.
* evaluate the correlation between Rheumatoid arthritis activity and subclinical structural changes of LA.
* determine the association of LA volume index and atrial fibrillation or HFpf in RA patients.
* apply Musculoskeletal Ultrasound detected synovitis to be correlated with cardiac function.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic progressive disease associated with systemic inflammation that affects mainly synovial joints leading to tissue destruction, disability and excess mortality (1). With a prevalence ranging from 0.4% to 1.3% of the population depending on both sex (women are affected two to three times more often than men), age (frequency of new RA diagnoses peaks in the sixth decade of life (2). RA has extra-articular manifestations that can impact multiple organ systems (3).

RA patients remain at higher cardiovascular risk compared to non-RA patients(4).Cardiovascular manifestations of RA include accelerated atherosclerosis, heart failure, pericarditis, myocarditis, endocarditis, rheumatoid nodules, and amyloidosis. Inflammation is an important mediator of endothelial dysfunction and is a key driver of cardiovascular risk and complications in patients with RA (3). The increased prevalence of atherosclerosis in RA seems to be associated with excess inflammatory burden and requires tailored screening strategies and management (1).

Heart structural abnormalities are more prevalent in RA-patients than in general population, such as pericarditis, increased left ventricle mass and valvular disease (5). Left atrial (LA) dilation predicts atrial fibrillation and congestive heart failure. It also increases the risk of developing thromboembolic events(6).

Echocardiography, including transthoracic two and three-dimensional echocardiography, Doppler imaging, myocardial deformation and transesophageal echo, is an established and widely available imaging technique for the identification of cardiovascular manifestations that are crucial for prognosis in rheumatic diseases. Echocardiography is also important for monitoring the impact of drug treatment on cardiac function, coronary microcirculatory function, valvular function and pulmonary artery pressures (7).

Left atrial volume index (LAVI), measured by two-dimensional (2D) echocardiography, is an accurate descriptor of LA volume, and is recommended in the latest guidelines for the diagnosis of heart failure with preserved ejection fraction (HFpEF) (8). At present, most previous studies focus solely on detecting the associations between baseline LAVI and clinical outcomes, with few attentions paid to the prognostic value of LAVI alteration for HFpEF.

Clinically, RA patients typically present with a recent onset of tender and swollen joints, morning joint stiffness, generalized sickness symptoms, as well as abnormal laboratory tests (2). The 28-joint disease activity score (DAS28) is a widely used measure to assess disease activity in rheumatoid arthritis (RA). The DAS28-P index, a derived proportion of the patient-reported components (joint tenderness and patient global assessment) within the DAS28, has been utilized as a discriminatory measure of non-inflammatory pain mechanisms in RA (9).

Both ultrasound and MRI have been recommended for diagnosing and monitoring disease activity in RA patients (10). Musculoskeletal ultrasound is widely used to identify structural change and assess therapeutic response in RA Ultrasound analysis (e.g., as high-resolution musculoskeletal ultrasound) of inflamed joints allows imaging of synovial proliferation by grayscale as well as both active inflammation and neoangiogenesis by power Doppler. In addition, ultrasound can identify bone erosions (11), as well as subclinical synovitis that may result in radiographic disease progression even if the patient is in apparent clinical remission (12).Due to these capabilities, ultrasound is widely used in clinical practice as well as in clinical trials for the diagnosis of RA and the monitoring of disease states (13).The advantages of ultrasound are its relatively low cost, wide availability, lack of contraindications, and non-invasive real-time imaging capabilities. Disadvantages are that ultrasound is considered an operator-dependent technology because of it being training-intensive in terms of both measurement and quality assessment (12).

While being a very sensitive diagnostic tool to detect e.g., synovial hypertrophy or pannus formation before the occurrence of bone erosion, routine usage of magnetic resonance imaging (MRI) techniques (preferably contrasted) in the diagnosis of RA is limited by cost factors and the limited capacity to image multiple joints in one measurement (2).

In our study, we will evaluate the LA function and dimensions, parallel to the evaluation of disease activity in RA patients, to detect possible association between disease activity and subclinical LA affection.

Sample size was calculated using epi info program. the following parameters were applied for observational cross sectional study. Population size 150 seek care at Assiut university hospital, proportion of left ventricular dysfunction among RA patients 59% (5) , design effect 1, and 95% confidence interval.

The minimum estimated Sample size was 108 RA patients. All participants will be subjected to the following: history taking and clinical examination, including Patients' data will be collected, included age at diagnosis, gender, residence, occupation, smoking and comorbidities, and duration , symptoms and signs of RA activity within the last 7 days. If articular activity is present, disease activity score-28 (DAS-28) will be calculated based on the number of swollen or tender joint count and will be applied to establish RA activity

Patients will be subjected to transthoracic echocardiography including, the following parameters will be measured:

* Left ventricular (LV) dimensions: end diastolic and systolic dimensions and LV ejection fraction (EF).
* Trans- mitral Doppler flow velocities including early (E) and late(A) diastolic velocities, E/A ratio.
* LA anteroposterior diameter measure from 2D parasternal long axis view targeted M-mode.
* LA superior-inferior and medio-lateral diameters measure from the apical 4 chamber view.
* LA volume included:
* Maximal LA volume measure at the end of systole just before mitral valve opening at the end of the T wave on ECG. Maximal LA volume is delivered from semi-automated tracing of the LA endometrium, starting the measurements in the frame with the largest atrial dimensions ,corresponding to ventricular end systole, just before the opening of the atrio-ventricular valves, in perpendicular apical long axis planes.
* Minimal LA volume will be measured at end diastole just at the closure of the mitral valve.
* Pre contractile LA volume ( LAV pre-A] measured at P-wave onset on ECG just before atrial contraction.

LA volume index (LAVI) will be obtained as the following: LA maximal volume will be obtained from apical four-chamber and two-chamber views at end-systole through the modified Simpson disc method, and then normalized to body surface area (BSA) to derive LAVI. This will be assessed according to ASE guidelines then the patients according to the measures will be into four different levels: normal (≤34 ml/m2), mild dysfunction (34-41 ml/m2), moderate dysfunction (42-48 ml/m2), and severe dysfunction (>48 ml/m2).

Laboratory investigations will be obtained

* Erythrocyte sedimentation rate (ESR).
* C reactive protein (CRP).
* Complete blood count (CBC).
* Lipid profile test

  * Musculoskeletal ultrasonography will be done: Ultrasound detected synovitis to be correlated with cardiac function.
  * X ray of Hands will be done.
  * Electrocardiogram (ECG) will be done. 2.4.1- Type of the study: Observational cross-sectional study 2.4. 2- Study Setting: rheumatology unit, Internal Medicine Department at Assiut University Hospitals.

2.4. 3- Study subjects:

1. Inclusion criteria:

   1. Patients with RA (aged >18 years and duration of RA disease >1 year) come to the rheumatology/ Internal medicine department or outpatient clinics at Assiut University Hospital.
   2. RA are diagnosed based on the ACR/EULAR 2010 rheumatoid arthritis classification criteria if a total score of ≥6 is needed to classify a patient as having definite RA.
2. Exclusion criteria:

   1- Patients with known history of atherosclerotic heart disease. 2- Patients with overlap syndrome. 3- Patients with hypothyroidism, Cushing's syndrome, anemia, and severe hepatic or renal dysfunction
3. Sample size Calculation:

   sample size was calculated using epi info program. the following parameters were applied for observational cross sectional study. Population size 150 seek care at Assiut university hospital, proportion of left ventricular dysfunction among RA patients 59% (5) , design effect 1, and 95% confidence interval.

   The minimum estimated Sample size was 108 RA patients. 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): A-History taking
   1. All participants will be subjected to the following: history taking and clinical examination, including Patients' data will be collected, included age at diagnosis, gender, residence, occupation, smoking and comorbidities, and duration , symptoms and signs of RA activity within the last 7 days. If articular activity is present, disease activity score-28 (DAS-28) will be calculated based on the number of swollen or tender joint count and will be applied to establish RA activity ,
   2. Type of treatment received, emphasizing current and former medications, B- Laboratory investigations • Erythrocyte sedimentation rate (ESR).

      • C reactive protein (CRP).

      • Complete blood count (CBC).

      • Lipid profile test.

      C- Other investigation:

      - Echocardiographic examination:

      Patients will be subjected to transthoracic echocardiography including, the following parameters will be measured:

      • Left ventricular (LV) dimensions: end diastolic and systolic dimensions and LV ejection fraction (EF).

      • Trans- mitral Doppler flow velocities including early (E) and late(A) diastolic velocities, E/A ratio.

      • LA anteroposterior diameter measure from 2D parasternal long axis view targeted M-mode.

      • LA superior-inferior and medio-lateral diameters measure from the apical 4 chamber view.

      • LA volume included:

      • Maximal LA volume measure at the end of systole just before mitral valve opening at the end of the T wave on ECG. Maximal LA volume is delivered from semi-automated tracing of the LA endometrium, starting the measurements in the frame with the largest atrial dimensions ,corresponding to ventricular end systole, just before the opening of the atrio-ventricular valves, in perpendicular apical long axis planes.
      * Minimal LA volume will be measured at end diastole just at the closure of the mitral valve.
      * Pre contractile LA volume ( LAV pre-A] measured at P-wave onset on ECG just before atrial contraction.

      LA volume index (LAVI) will be obtained as the following: LA maximal volume will be obtained from apical four-chamber and two-chamber views at end-systole through the modified Simpson disc method, and then normalized to body surface area (BSA) to derive LAVI. This will be assessed according to ASE guidelines then the patients according to the measures will be into four different levels: normal (≤34 ml/m2), mild dysfunction (34-41 ml/m2), moderate dysfunction (42-48 ml/m2), and severe dysfunction (>48 ml/m2).

      - Musculoskeletal ultrasonography : Ultrasound detected synovitis to be correlated with cardiac function.

      - X ray of Hands.

      - Electrocardiogram (ECG). 2.4.5 -Research outcome measures:

      Primary (main):

      • Detect echocardiographic abnormalities in patients with rheumatoid arthritis.
      * Detect subclinical echocardiographic changes of the LA (dimensions and function) in patients with rheumatoid arthritis..
      * Evaluate the correlation between Rheumatoid arthritis and increased heart failure risk..

      Secondary outcome (Subsidiary) :
      * Describe concurrent systemic comorbidities, rheumatologic clinical activity, serologic markers of rheumatoid arthritis, and inflammatory activity.
      * Evaluation of the LA function and dimensions, parallel to the evaluation of disease activity in RA patients, to detect possible association between disease activity and subclinical LA affection.

      Data management and analysis:

      Data collection: The collected data will be revised, coded, tabulated and introduced to a PC.

      Computer software IBM_SPSS. Statistical Package for Social Science. Ver.21. Standard version. Copyright © SPSS Inc., 2011-2012. NY, USA. 2012.

      Statistical tests Data will be presented, and suitable analysis will be done according to the type of data obtained for each parameter.

i.Descriptive statistics:

1.Description of qualitative variables is done by frequency and percentage. 2.Description of quantitative variables is in the form of mean and SD. ii.Analytic statistics:

1. χ2-test and Fisher's exact test are used for comparison of qualitative variables with each other.
2. Comparison between quantitative variables is carried out using Student's t-test of two independent samples.
3. For comparison of more than two quantitative groups, analysis of variance F-test is used for categorical data.
4. Significance level (P) is expressed as follows: P value greater than 0.05 is not significant, P value less than 0.05 is significant, and P value less than 0.001 is highly significant.
5. Pearson's correlation coefficient is used to calculate the correlation between quantitative variables.

Spearman's coefficient is calculated to determine the relationships between non parametric quantitative variables

ELIGIBILITY:
Inclusion Criteria:

- 1- Patients with RA (aged >18 years and duration of RA disease >1 year) come to the rheumatology/ Internal medicine department or outpatient clinics at Assiut University Hospital.

2-RA are diagnosed based on the ACR/EULAR 2010 rheumatoid arthritis classification criteria if a total score of ≥6 is needed to classify a patient as having definite RA

Exclusion Criteria:

1. Patients with known history of atherosclerotic heart disease.
2. Patients with overlap syndrome.
3. Patients with hypothyroidism, Cushing's syndrome, anemia, and severe hepatic or renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be from rheumatology unit, Internal Medicine Department at Assiut University Hospitals and its outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
• Detect echocardiographic abnormalities in patients with rheumatoid arthritis | 4 hours
  * Detect echocardiographic abnormalities in patients with rheumatoid arthritis.
  * Detect subclinical echocardiographic changes of the LA (dimensions and function) in patients with rheumatoid arthritis..
  * Evaluate the correlation between Rheumatoid arthritis and increased heart failure risk.
perform musculoskeletal Ultrasound detected synovitis to be correlated with cardiac function. | 4 hours

SECONDARY OUTCOMES:
• Evaluation of the LA function and dimensions, parallel to the evaluation of disease activity in RA patients, to detect possible association between disease activity and subclinical LA affection. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Salwa salah elgendi, MD, Study Director — assuit univeristy hospitals; Taghreed sayed Meshref, MD, Study Director — assuit univeristy hospitals; Abdelhafeez Mohmoud Moshrif, MD, Study Director — Al-Azhar faculty of medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erre GL, Chessa I, Bassu S, Cavagna L, Carru C, Pintus G, Giordo R, Mangoni AA, Damiano Sanna G, Zinellu A. Association between ischemia-modified albumin (IMA) and peripheral endothelial dysfunction in rheumatoid arthritis patients. Sci Rep. 2024 Feb 17;14(1):3964. doi: 10.1038/s41598-024-54641-5. PMID 38368495
- [Background] Takase-Minegishi K, Horita N, Kobayashi K, Yoshimi R, Kirino Y, Ohno S, Kaneko T, Nakajima H, Wakefield RJ, Emery P. Diagnostic test accuracy of ultrasound for synovitis in rheumatoid arthritis: systematic review and meta-analysis. Rheumatology (Oxford). 2018 Jan 1;57(1):49-58. doi: 10.1093/rheumatology/kex036. PMID 28340066
- [Background] Wang YW, Chen JF, Ko CH, Cheng TT, Chiu WC, Yu SF, Hsu CY, Chen YC. Factors associated with subclinical inflammation of wrist joints in rheumatoid arthritis patients with low or no disease activity- a RA ultrasound registry study. BMC Musculoskelet Disord. 2023 May 30;24(1):438. doi: 10.1186/s12891-023-06521-8. PMID 37254118
- [Background] Chen CC, Chen DY. The Clinical Utility of Musculoskeletal Ultrasound for Disease Activity Evaluation and Therapeutic Response Prediction in Rheumatoid Arthritis Patients: A Narrative Review. J Med Ultrasound. 2023 Nov 10;31(4):275-281. doi: 10.4103/jmu.jmu_126_22. eCollection 2023 Oct-Dec. PMID 38264607
- [Background] Sudol-Szopinska I, Jans L, Teh J. Rheumatoid arthritis: what do MRI and ultrasound show. J Ultrason. 2017 Mar;17(68):5-16. doi: 10.15557/JoU.2017.0001. Epub 2017 Mar 31. PMID 28439423
- [Background] Pisaniello HL, Whittle SL, Lester S, Menz F, Metcalf R, McWilliams L, Hill CL, Proudman S. Using the derived 28-joint disease activity score patient-reported components (DAS28-P) index as a discriminatory measure of response to disease-modifying anti-rheumatic drug therapy in early rheumatoid arthritis. BMC Rheumatol. 2022 Nov 15;6(1):67. doi: 10.1186/s41927-022-00299-3. PMID 36376988
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Böhm M, et al. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC) With the special contribution of the Heart Failure Association (HFA) of the ESC. European heart journal. 2021;42(36):3599-72
- [Background] Makavos G, Varoudi M, Papangelopoulou K, Kapniari E, Plotas P, Ikonomidis I, Papadavid E. Echocardiography in Autoimmune Rheumatic Diseases for Diagnosis and Prognosis of Cardiovascular Complications. Medicina (Kaunas). 2020 Sep 1;56(9):445. doi: 10.3390/medicina56090445. PMID 32883041
- [Background] Foglieni C, Rusconi R, Mantione ME, Fragasso G, Alfieri O, Maisano F. Early left atrial tissue features in patients with chronic mitral regurgitation and sinus rhythm: Alterations of not remodeled left atria. Int J Cardiol. 2016 Sep 15;219:433-8. doi: 10.1016/j.ijcard.2016.06.047. Epub 2016 Jun 15. PMID 27372606
- [Background] Corrao S, Messina S, Pistone G, Calvo L, Scaglione R, Licata G. Heart involvement in rheumatoid arthritis: systematic review and meta-analysis. Int J Cardiol. 2013 Sep 1;167(5):2031-8. doi: 10.1016/j.ijcard.2012.05.057. Epub 2012 Jun 15. PMID 22703938
- [Background] Park E, Bathon J. Cardiovascular complications of rheumatoid arthritis. Curr Opin Rheumatol. 2024 May 1;36(3):209-216. doi: 10.1097/BOR.0000000000001004. Epub 2024 Feb 9. PMID 38334476
- [Background] Sanghavi N, Ingrassia JP, Korem S, Ash J, Pan S, Wasserman A. Cardiovascular Manifestations in Rheumatoid Arthritis. Cardiol Rev. 2024 Mar-Apr 01;32(2):146-152. doi: 10.1097/CRD.0000000000000486. Epub 2022 Nov 21. PMID 36729119
- [Background] Lin YJ, Anzaghe M, Schulke S. Update on the Pathomechanism, Diagnosis, and Treatment Options for Rheumatoid Arthritis. Cells. 2020 Apr 3;9(4):880. doi: 10.3390/cells9040880. PMID 32260219
- See also: Related Info — https://www.nature.com/articles/s41598-021-00657-0